CLINICAL TRIAL: NCT02858518
Title: Risk of Bleeding and Anticoagulation in Atrial Fibrillation: What Predictive Criterion Used?
Acronym: PREDIC-AGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408020; 2014-A01664-43 (Other: ANSM)
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation; Gerontology
Keywords: anticoagulant
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — classical blood sample : NFS, ionograms, CRP, TSH, albumin, vitamin D, Calcium and coagulation factors + tube for genetic study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with atrial fibrillation with anticoagulant treatment
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — scales : HEMORR2HAGES (hepatics diseases, alcoholism, cancer, thrombocytopenia, anemia and antecedent...), HAS-Bled (arterial hypertension, renal function, liver function, cerebrovascular accident...), ATRIA (anemia, serious kidney diseases, hypertension, antecedent...), Shireman (gender, age, hemorrhage, diabetes, anemia...), Charlson (age, cardiovascular disease, lung disease, neurological disease, endocrinal disease, nephrology, liver disease, gastroenterology, cancer) and standardised geriatric assessment (comorbidities, cognition, mobility, pain, nutrition, living environment...)

SUMMARY:
Atrial fibrillation (AF) is a rhythmic cardiac activity disorder disturbing hemodynamic blood flow. It is a public health problem with 600,000 to 1 million people involved in France which 2/3 are aged over 75 years. a FA untreated exposes the patient to a significant risk of embolism responsible for a rate stroke (stroke) ischemic estimated at 85%. The anticoagulant standard treatment helps prevent the occurrence of this complication.

However, oral anticoagulation also exposes patients to an increased risk of bleeding. The bleeding risk can be assessed using scales: several being proposed (HEMORR2HAGES, HAS-BLED, ATRIA and scores Shireman and Charlson ...).

moreover, in geriatric hospital care, every patient has a "standardized geriatric assessment" to assess and quantify functional capacity, autonomy, cognitive abilities, nutritional status, psychological state and its environment social.

Thus, the objective of the investigators study was to determine the frequency of each item of each bleeding risk assessment score and geriatric assessment in patients 80 and older hospitalized geriatric ward in the department and with anticoagulant.

ELIGIBILITY:
Inclusion Criteria:

* hospitalisation in geriatric unit
* Atrial fibrillation treated by anticoagulant treatment (AVK or oral anticoagulation)
* signed inform consent

Exclusion Criteria:

* estimated lifetime less than 6 months
* under guardianship or curatorship
* without support person

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients seniors with atrial fibrillation with anticoagulant treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
scale : HEMORR2HAGES | at baseline
  hepatics diseases, alcoholism, cancer, thrombocytopenia, anemia and antecedent...
scale : HAS-Bled | at baseline
  arterial hypertension, renal function, liver function, cerebrovascular accident...
scale : ATRIA | at baseline
  anemia, serious kidney diseases, hypertension, antecedent...
scale : shireman | at baseline
  gender, age, hemorrhage, diabetes, anemia...
scale charlson | at baseline
  age, cardiovascular disease, lung disease, neurological disease, endocrinal disease, nephrology, liver disease, gastroenterology, cancer
scale : standardised geriatric assessment | at baseline
  comorbidities, cognition, mobility, pain, nutrition, living environment...

SECONDARY OUTCOMES:
Occurrence of major bleeding event or not major | at baseline and 6 months
genotyping | at baseline
  CYP2C9
genotyping | at baseline
  VKCRC1

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CRAWFORD-ACHOUR, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (5):
- France (5):
  - CH de FEURS, Feurs
  - CH de FIRMINY, Firminy
  - CH de ROANNE, Roanne
  - CH de SAINT-CHAMOND, Saint-Chamond
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No